CLINICAL TRIAL: NCT00597051
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled, Cross-Over, Multi-Centre Study of the Pharmacokinetics and Tolerability of 3 Different Doses of ARD-0403 in Testosterone Deficient Men
Brief Title: Study of 3 Doses of ARD-0403 in Testosterone Deficient Men
Acronym: ARD-0403-001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ardana Bioscience Ltd (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ARD-0403-001
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2008-01-17 (Estimated); Status verified 2008-01

CONDITIONS: Hypogonadism
MeSH Terms: conditions — Hypogonadism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ARD-0403

SUMMARY:
The purpose of this study is to determine which dose, if any, results in testosterone levels within the normal range for men.

ELIGIBILITY:
Inclusion Criteria:

* Testosterone deficiency
* Normal BMI

Exclusion Criteria:

* Previous treatment with testosterone replacement therapy within 4 weeks
* Moderate-severe benign prostatic hypertrophy, or prostatic cancer
* Haematocrit >50%

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-10; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Mokhort, MD, Principal Investigator — Republican Endocrinology Center Hospital, Minsk, Republic of Belarus
Locations (1):
- Republican Endocrinology Center Hospital, Minsk, Belarus